CLINICAL TRIAL: NCT01551433
Title: A Prospective Trial to Evaluate Whether Variations in Tissue Oxygenation Are Associated With Anastomotic Leak Rates After an Ivor Lewis Esophagectomy
Brief Title: Tissue Oxygenation Are Associated With Anastomotic Leak Rates After an Ivor Lewis Esophagectomy
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 11-192
Record Dates: First submitted 2012-03-01; First posted 2012-03-12 (Estimated); Last update posted 2016-08-18 (Estimated); Status verified 2016-08

CONDITIONS: Esophageal Cancer
Keywords: esophagectomy; ESOPHAGUS; Wipox instrument; Tissue Oxygenation; Anastomotic Leak; 11-192
MeSH Terms: conditions — Esophageal Neoplasms; Anastomotic Leak | interventions — Diathermy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Pts scheduled for Ivor Lewis esophagectomy: During the operation, once the gastric conduit has been mobilized and positioned, and once the anastomotic site has been identified by the surgeon, the assigned RSA will provide the Wipox instrument to the fellow (the primary surgeon will be blinded to the result) who will then obtain one measurement from the anastomotic site.
  Interventions: Device: wireless pulse oximeter (Wipox)

INTERVENTIONS:
Device: wireless pulse oximeter (Wipox) — In addition to the one Wipox measurement at the planned anastomotic site, the RSA will collect the systemic pulse oximeter reading, blood pressure, and heart rate at the time of the Wipox measurement. These measurements will be obtained as both internal controls of the accuracy of the Wipox (matching the Wipox pulse rate with the patient's), as well as additional variables to control for when assessing factors which might contribute to oxygen saturation at the anastomotic site. Pre-operative demographic information will be collected. This will include age, sex, any co-morbidities (cardiac, diabetes, respiratory), and use of pre-operative chemotherapy or chemo-radiotherapy.
  Other Names: Post-operatively, all complications will be recorded and graded by the RSA.; Anastomotic leaks present either symptomatically or asymptomatically. An; asymptomatic leak is only detected on the routine post-operative esophagram on; post-operative days 5-7, and is isusally described as a 'contained leak'. A; symptomatic leak is usually becomes evident due to clinical symptoms such as a; fever, leukocutosis, or enteric contents in the periesophageal drains.

SUMMARY:
The purpose of this study is to test whether after an Ivor Lewis esophagectomy (the removal of a portion of the stomach and esophagus with re-attachment) there is an association between the intraoperative level of oxygen at the site where the esophagus is re-attached to the stomach (measured using the Wipox), and the incidence of a disruption at the site of the attachment after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are scheduled to undergo an open or a minimally invasive Ivor Lewis esophagectomy
* > or = to 21 years of age

Exclusion Criteria:

* Patients who are not candidates for an esophagectomy as determined by the treating surgeon

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The Thoracic Surgery clinics
Sampling Method: Non-Probability Sample
Enrollment: 166 (Actual)
Dates: Start 2012-02; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
association between tissue oxygenation (measured using the Wipox) at the anastomotic site and the incidence of anastomotic leak after an Ivor Lewis esophagectomy. | 2 years
  The primary objective of this observational study is to determine whether in patients undergoing Ivor Lewis esophagectomy, low levels of tissue oxygenation at the anastomotic site are associated with increased risk of anastomotic leak (AL).

SECONDARY OUTCOMES:
To correlate various demographic | 2 years
  (age, co-morbidities, smoking history) and clinical variables (pre-operative therapy, intra-operative blood pressure and systemic oxygen saturation) with tissue oxygenation at the anastomotic site. Spearman rank correlation (for continuous variables) and Wilcoxon rank sum test (for categorical variables) will be used to test these associations.
To correlate anastomotic site tissue oxygenation with the postdischarge incidence of stricture | 2 years
  the association between anastomotic site tissue oxygenation and the incidence of post-discharge stricture observed during the 6 months following surgery will be assessed using Wilcoxon rank sum test (with O2 levels on a continuous scale) and Fisher exact test.
To correlate clinical variables | 2 years
  (age, co-morbidities, smoking history) and clinical variables (pre-operative therapy, intra-operative blood pressure and systemic oxygen saturation) with tissue oxygenation at the anastomotic site. Spearman rank correlation (for continuous variables) and Wilcoxon rank sum test (for categorical variables) will be used to test these associations.

CONTACTS AND LOCATIONS:
Overall Officials: Prasad Adusumilli, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/